CLINICAL TRIAL: NCT00450515
Title: Phase II Trial of Vinfluinine and Capecitabine in Previously Treated Metastatic Breast Cancer
Brief Title: Vinflunine and Capecitabine in Treating Patients With Previously Treated Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was dropped prior to opening.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0632; NCI-2011-01743 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000536545 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Capecitabine; vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vinflunine + capecitabine (Experimental): Patients receive vinflunine IV over 20 minutes on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline, every other course, and at the completion of study treatment.
  After completion of study treatment, patients are followed periodically for up to 5 years.
  Interventions: Drug: capecitabine; Drug: vinflunine

INTERVENTIONS:
Drug: capecitabine
Drug: vinflunine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinflunine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vinflunine together with capecitabine works in treating patients with previously treated metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the tumor response rate in patients with previously treated metastatic breast cancer treated with vinflunine and capecitabine.

Secondary

* Describe the adverse event profile of this regimen in these patients.
* Determine the progression-free survival of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the duration of response in patients treated with this regimen.
* Determine the time to treatment failure in patients treated with this regimen.
* Describe the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive vinflunine IV over 20 minutes on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every other course, and at the completion of study treatment.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer meeting the following criteria:

  * Metastatic disease
  * Previously treated with 1-2 chemotherapy regimens for metastatic disease
* Measurable disease, defined as ≥ 1 measurable lesion ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan

  * No nonmeasurable disease, including any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* Must have received ≥ 1 prior trastuzumab (Herceptin®)-containing regimen (unless there is a contraindication) if tumor is HER2 positive (3+ by immunohistochemistry or amplified by fluorescent in situ hybridization [FISH])
* No CNS metastasis unless controlled by prior surgery and/or radiotherapy

  * "Controlled" is defined as ≥ 2 months of no symptoms or evidence of progression
* Currently enrolled on clinical trial QOL N0392
* Hormone receptor status not specified

  * Hormone-positive tumor must meet at least 1 of the following criteria:

    * Tumor refractory to hormonal therapy
    * Heavy visceral tumor burden that requires chemotherapy for better and faster control of metastatic disease
    * Relapsed disease during adjuvant hormonal therapy and failed first-line chemotherapy
    * Not treated with hormonal therapy because of side effects or adverse events

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 8.0 g/dL
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase (AP), AST, and ALT must meet 1 of the following criteria:

  * AP normal AND AST and ALT ≤ 5 times ULN
  * AP ≤ 2.5 times ULN AND AST and ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST and ALT normal
* Creatinine clearance ≥ 30 mL/min
* Serum sodium normal
* Not pregnant or nursing

  * No nursing during and for 30 days after completion of study therapy
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study therapy
* No history of allergy or hypersensitivity to drug product excipients or to agents chemically similar to vinflunine and/or capecitabine
* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No known hypersensitivity to fluorouracil
* No known dihydropyrimidine dehydrogenase deficiency
* No active, unresolved infection
* No New York Heart Association class III-IV cardiovascular disease, unstable angina, myocardial infarction within the past 6 months, or poorly controlled hypertension
* No preexisting neuropathy ≥ grade 2
* No concurrent serious medical condition that would preclude study treatment
* No other stage III or IV invasive cancer within the past 3 years
* No lack of physical integrity of the upper gastrointestinal tract, clinically significant malabsorption syndrome, or inability to take oral medication
* Ability to complete questionnaires alone or with assistance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior unlimited hormonal therapy allowed in the neoadjuvant, adjuvant, or metastatic setting
* No major surgery, chemotherapy, or immunologic therapy within the past 4 weeks
* No radiotherapy within the past 4 weeks, except if to a nontarget lesion only

  * Prior radiotherapy to a target lesion is allowed if there has been clear progression of the lesion since radiotherapy was completed
  * If patient received single-dose radiotherapy or palliation to a nontarget lesion only, the patient may immediately proceed to study registration without waiting 4 weeks
* No prior fluoropyrimidines, including capecitabine, or vinca alkaloids (e.g., vinorelbine, vinblastine, vincristine, or vindesine) for metastatic breast cancer
* No prior radiotherapy to > 30% of bone marrow-containing areas
* No cimetidine, allopurinol, sorivudine, or brivudine within the past 2 weeks
* No ketoconazole, itraconazole, ritonavir, amprenavir, or indinavir within the past 2 weeks
* No concurrent treatment in another clinical trial in which investigational procedures are performed or investigational therapies are administered
* No concurrent trastuzumab (Herceptin®)
* No concurrent hormonal therapy
* No concurrent interleukin-11
* No other concurrent chemotherapeutic agents, biologic agents, or radiotherapy
* No concurrent administration of any of the following:

  * Cimetidine
  * Allopurinol
  * Sorivudine
  * Brivudine
  * Ketoconazole
  * Itraconazole
  * Ritonavir
  * Amprenavir
  * Indinavir
* Warfarin allowed if patient is on a stable dose and has an INR < 3.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response | Up to 10 years

SECONDARY OUTCOMES:
Adverse event profile | Up to 10 years
Progression-free survival | Up to 10 years
Overall survival | Up to 10 years
Duration of response | Up to 10 years
Time to treatment failure | Up to 10 years
Quality of life | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Moreno, MD, Study Chair — Mayo Clinic